CLINICAL TRIAL: NCT00000288
Title: Role of Metabolites in Nicotine Dependence (2)
Brief Title: Role of Metabolites in Nicotine Dependence (2) - 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-5; P50-09259-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Drug: Cotinine fumarate

SUMMARY:
The purpose of this study is to determine the effects of varying doses of cotinine on cigarette self-administration.

DETAILED DESCRIPTION:
Previous studies have shown that cotinine, a metabolite of nicotine, antagonizes some of the effects of nicotine. One study showed that nicotine eliminates some of the beneficial effects of the nicotine patch in reducing withdrawal symptoms. The purpose of this study was to examine the effects of cotinine. The results generally showed no effects on self-administration of cigarettes, although higher serum nicotine levels were observed on the highest doses of cotinine compared to placebo or lower doses of cotinine.

ELIGIBILITY:
Inclusion Criteria:

Male/Female subjects ages 21-45 yrs. inclusive, with a smoking history of at least 1 pack of cigarettes daily for at least 1 year. Subject must be in good health as verified by medical history, screening examination, and screening laboratory tests. Subject must provide written informed consent to participate in the study and be motivated to stop smoking for a short term.

Exclusion Criteria:

History of myocardial infarction, angina pectoris, sustained or episodic cardiac arrhythmias, symptomatic peripheral vascular disease, peptic ulcer disease or any other medical condition which the physician or investigator deems inappropriate for participation. Insulin-dependent diabetes. Pregnant or lactating, or not using adequate birth control methods. Requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history). Chronic use of systemic steroids or antihistamines. Skin sensitivity which would preclude use of a transdermal system. Abuse of alcohol or any other recreational or prescription drug. Use of any other tobacco products including smokeless tobacco and nicotine products. Previous use of transdermal nicotine system. Inability to fulfill all scheduled visits and examination procedures throughout the study period.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-12; Study Completion 2002-12

PRIMARY OUTCOMES:
Subjective effects
Physiological effects
Behavioral
Subjective

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Presented at Society for Research on Nicotine and Tobacco Scientific Meeting, 1997 and Psychopharmacology 1998. Presented at Society for Research on Nicotine and Tobacco Scientific Meeting, 1997.